CLINICAL TRIAL: NCT06681844
Title: Prediction of the Tooth Wear Index Based on a Dataset of Dental Shapes:a Retrospective Study
Brief Title: Predict Tooth Wear
Acronym: PREDITOOTH
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1046
Record Dates: First submitted 2023-11-10; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Prediction of Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- all mature teeth presenting a tooth wear intact or presenting a tooth wear altered: Scaling of the tooth before scanning by the operator Evaluation of the tooh wear index 0 or 1 (by 2 calibrated experts )
  Interventions: Other: Tooth Shape assessed using an intraoral scanner one after avulsion

INTERVENTIONS:
Other: Tooth Shape assessed using an intraoral scanner one after avulsion — * Tooth Shape assessed using an intraoral scanner one after avulsion and stored as StereoLithography (STL) file
  * Age, gender, reason of avulsion, type of tooth taken from the database and stored in a google sheet

SUMMARY:
Tooth wear, resulting from gradual loss of dental hard tissue due to mechanical and chemical factors, impacts tooth structure, texture, and function. It affects quality of life, with varying prevalence (26.9% to 90.0%), and is traditionally detected visually during check-ups, often at advanced stages. Monitoring alterations in tooth shape via intraoral scanners aids early detection, but restoration remains challenging. Prevention through early detection is vital, as patients may not fully comprehend tooth structure loss until visible. Recently, statistical shape analysis (SSA) used to learn the tooth anatomy and define a reference shape (biogeneric tooth) using. However, assuring landmark consistency is challenging mostly due to biases of the operator. Recently, a robust method called MEG-IsoQuad offered automated, isotopological remeshing. Combining this with SSA holds promise for diagnostic and simulation purposes. This study aims to assess the reliability of a remeshing-SSA approach for altered and intact premolar analysis and compare machine learning algorithms for simulating the shape of the initially intact tooth or future altered one.

The clinical perspective of the current work offers possibilities to:

* Prevent future tooth wear by detecting it at an early stage; and communicate better to the patient by presenting him/her potential future altered teeth
* Simulate the adapted reconstruction for the altered tooth by simulating the initially intact one

ELIGIBILITY:
Inclusion Criteria:

* teeth avulsed presenting a tooth wear index between 0 and 3
* mature incisor, canine, premolar or molars (1st and 2nd only)

Exclusion Criteria:

* teeth avulsed presenting a tooth wear index over 3 (or presenting an oral rehabilitation representative of a similar wear)
* immature teeth or teeth without root edification
* wisdom teeth

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Avulsed teeth at the Oral Surgery Departement of the Lyon Dental University Hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of the tooth wear index based on a dataset of dental shapes:a retrospective study | only once
  Four machine learning (ML) algorithms: a linear discriminant analysis (LDA) a support vector machine (SVM), a random forest (RM) and a gradient boosting machine (GBM) will be used to predict the tooth type and the alteration of the anatomy. The data set will be split into a 60/40 train and holdout test data set and models will be three-fold cross validated. Model performances will be evaluated in confusion matrices leading to define precision, recall, F1 score and accuracy.

CONTACTS AND LOCATIONS:
Locations (5):
- Indiana University Hospital, Indianapolis, Indiana, United States
- KU Leuven University Hospital, Leuven, Belgium
- Lyon Dental Hospital, Lyon, France
- King George Medical University, Lucknow, India
- Tel Aviv Universi, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No